CLINICAL TRIAL: NCT01526239
Title: Patient-Reminder Results in Patient-Initiated Promoting Colorectal Cancer Screening Via Colonoscopy
Brief Title: Reminding Patients of the Important of Colorectal Cancer Screening Results in Patient-Initiated Promoting Colorectal Cancer Screening Via Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 14225
Record Dates: First submitted 2012-01-03; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Colon Cancer
Keywords: Colorectal cancer screening; colon cancer screening; colonoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention consisted of a pamphlet about the benefit of CRC-S, given to patients prior to their PCP visit and a reminder note about CRC screening to be given to their physician during the encounter.
  Interventions: Other: Colorectal cancer screening pamphlet
- Control group (No Intervention): Control group will not receive the pamphlet regarding colorectal cancers.

INTERVENTIONS:
Other: Colorectal cancer screening pamphlet — Colorectal cancer screening pamphlet
  Arms: Intervention group

SUMMARY:
Colorectal cancer is the third most common cancer diagnosed and third leading cause of cancer-related deaths in the United States for both men and women. The American Cancer Society (ACS) estimates about 108,070 new cases of colon cancer and 40,740 new cases of rectal cancer will be diagnosed, and about 49,960 deaths will occur as a result of this devastating disease in 2008. Over the last 20 years, the death rate for this cancer has been dropping as a result of screening and early detection of cancer. In 2007, ACS reported that early-stage colorectal cancer had a survival rate close to 80%, and up to 9,632 deaths could be prevented each year if eligible patients received screening when necessary. However, despite the proven efficacy of colorectal cancer (CRC) screening, only about 50% of eligible US patients are currently being screened.

Specific Aims

The central hypothesis of this proposal is that patient-initiated prompting of primary care physicians of the patient's interest in screening will increase referrals for CRC screening. The following three areas will be investigated during this research:

1. To determine whether a communication tool provided to patients will initiate a conversation with their primary care physicians about CRC screening, especially via colonoscopy.
2. To determine whether this tool will impact referral patterns for screening, especially, although not primarily, among poor and underserved populations.
3. To determine whether differences exist in regard to patient-physician communication patterns about screening among residents and faculties in the fields of internal medicine and family practice clinics.

At the close of the investigators study, the investigators wish to organize quantifiable data demonstrating how patient-initiated prompting of primary care physicians for CRC screening increases early detection and decreases potential mortality from colorectal cancer. This data will inform a second, larger study to pursue the questions surrounding patient-initiated prompting in

ELIGIBILITY:
Inclusion Criteria:

* All patient age older than 50, exception for African American age 45 and older

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Communication with primary care physicians about CRC screening | 2 years
  The central hypothesis of this proposal is that patient-initiated prompting of primary care physicians of the patient's interest in screening will increase referrals for CRC screening.

CONTACTS AND LOCATIONS:
Locations (1):
- OUHSC HSC, GI department, Oklahoma City, Oklahoma, United States